CLINICAL TRIAL: NCT01059084
Title: An Open-label Trial of the Effect of Valacyclovir on Plasma HIV-1 Levels Among HIV-1 Seropositive and HSV-1/2 Seronegative Persons
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to enroll any participants into this study.
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Anna Wald, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 37304-B
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Valacyclovir; Valtrex®
MeSH Terms: conditions — HIV Infections | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Valacyclovir — 1000 mg tid

SUMMARY:
The purpose of this study is to look at the effect of daily herpes medication, valacyclovir, on HIV levels in the blood in persons who are HIV positive and do not have oral or genital herpes.

DETAILED DESCRIPTION:
The purpose of this study is to look at the effect of daily herpes medication, valacyclovir on HIV levels in the blood in persons who do not have genital herpes. This will help better understand the effect that valacyclovir plays in the spread of HIV and the potential role for HIV treatment in decreasing the HIV spread.

A total of 20 individuals who are HIV-1 seropositive and HSV-1/2 seronegative will be recruited for the study. Participants must not be on antiretroviral therapy and must not be planning to initiate HIV antiretroviral therapy during the study.

Participants will be asked to come to the clinic for a total of 16 visits over the course of 10 weeks. Participants will receive valacyclovir 1000 mg three times daily for 6 weeks. During the first week, participants will return to the clinic for a total of 2 visits and will provide plasma samples for baseline HIV-1 levels. During the second week, participants will return to the clinic for a total 5 visits. At Visit 3, participants will be provided the study medication. After drug initiation, participants will be asked to return to the clinic within 6 hours and then again at Day 1, 2, and 3 post first dose. During weeks 3-8, participants will be instructed to take valacyclovir and return to the clinic for one follow-up visit each week to provide plasma samples for HIV-1 detection.

Participants will be asked to return to the clinic for 3 follow-up visits after study drug discontinuation to provide plasma samples for HIV-1 detection.

Participants will be asked to complete a daily symptom and medication diary. All supplies and study medical will be provided.

This is an outpatient study.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* HIV-1 seropositive
* CD4 count>250 cell/mm3
* Detectable HIV-1 plasma viral load
* HSV-1 & 2 seronegative.
* Not on HIV antiretroviral therapy or planning to initiate antiretroviral therapy during the study period.
* Not intending to move out of the area for duration of study participation
* Willing and able to provide independent written informed consent.
* Willing and able to undergo clinical evaluations.
* Willing and able to take study drug as directed.
* Willing and able to adhere to follow-up schedule

Exclusion Criteria:

* Known history of adverse reaction to acyclovir, valacyclovir, or famciclovir.
* Use of ganciclovir, foscarnet, or cidofovir
* History of evidence of CMV disease
* Known medical history of seizures
* Known renal insufficiency, defined as serum creatine >1.5 mg/dl
* AST or ALT >3times upper limit of normal
* Hematocrit <30%
* Neutropenia, defined as absolute neutrophil count <1000
* Thrombocytopenia, defined as platelet count <75,000
* History of thrombotic microangiopathy
* For women, pregnancy as confirmed by a urine pregnancy test
* Any other condition which, in the opinion of the principal investigator, may compromise the ability to follow study procedures and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate plasma HIV-1 levels after treatment with valacyclovir compared to baseline HIV-1 levels before treatment. | Weeks (1-10)

SECONDARY OUTCOMES:
To determine frequency of reverse transcriptase drug resistant mutations in HIV-1 after exposure to valacyclovir | Weeks 7 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, MD, MPH, Principal Investigator — University of Washington